CLINICAL TRIAL: NCT02066584
Title: The Influence of Different Concentrations of Glucose in Culture Media on In Vitro Fertilization Outcome of Sibling Oocytes
Brief Title: The Influence of Different Concentrations of Glucose in Culture Media on In Vitro Fertilization (IVF) Outcome of Sibling Oocytes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0011-14HYMC
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
Keywords: sibling oocytes; glucose; culture media
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Universal IVF Medium: An oocyte culture medium containing 5.55 Mm glucose (Origio, Medi-Cult)
  Interventions: Other: Sibling oocyte incubation
- ISM1 Medium: An oocyte culture medium containing 1mM glucose ((Origio, MediCult)
  Interventions: Other: Sibling oocyte incubation
- P1 Medium: An oocyte culture medium containing no glucose (Irvine)
  Interventions: Other: Sibling oocyte incubation
- ECM Medium: An oocyte culture medium containing 0.5mM glucose (Irvine)
  Interventions: Other: Sibling oocyte incubation

INTERVENTIONS:
Other: Sibling oocyte incubation

SUMMARY:
The importance of glucose in culture media on fertilization and embryo development is still controversial. Although it has been reported that glucose is essential for fertilization process and biosynthesis of membrane lipid and nucleic acids, comparatively high levels of glucose in culture media may cause developmental arrest of cleavage stage embryos. The aim of this retrospective study is to examine whether exposure of sibling oocytes to different concentrations of glucose in culture media has any further effect on IVF outcome.

DETAILED DESCRIPTION:
This retrospective study will include data from either standard IVF or Intracytoplasmic Sperm Injection (ICSI) cycles, in which sibling oocytes were equally divided and incubated separately in one of the following pairs of culture media:

1. Universal IVF medium vs. ISM1 medium ( Origio, Medi-Cult)
2. P1 medium vs. ECM medium (Irvine).

Fertilization rate,as well as embryo cleavage rate and morphology will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Sibling oocytes from cycles where at least 4 oocytes were retrieved

Exclusion Criteria:

* Less than 4 oocytes retrieved
* Partner has undergone testicular sperm extraction (TESE)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sibling oocytes retrieved from women who have undergone IVF treatment in our IVF unit.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Fertilization Rate | 2 years
  Fertilization rates will be retrospectively compared according to culture media in which sibling oocytes were incubated

SECONDARY OUTCOMES:
Embryo Quality | 2 years
  Embryo quality and developmental rate will be retrospectively compared according to culture media in which sibling oocytes were incubated

CONTACTS AND LOCATIONS:
Overall Officials: Medeia Michaelo, PhD, Principal Investigator — Hellel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel